CLINICAL TRIAL: NCT04907370
Title: Toripalimab Combined With Induction Chemotherapy Followed by Radiotherapy Alone or Concurrent Chemoradiotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma: A Phase 3, Multi-center, Randomized Controlled Trial
Brief Title: PD-1 Blockade Combined With De-intensified Chemoradiotherapy Sparing Concurrent Cisplatin in Nasopharyngeal Carcinoma
Acronym: DIAMOND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Vice President of SYSUCC, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS001-ISS-CO291
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Immune checkpoint inhibitor; Radiotherapy; Concurrent cisplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Immune Checkpoint Inhibitors; Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab Combined with Induction Chemotherapy Followed by Radiotherapy Alone (Experimental): All participants will receive induction chemotherapy (IC; every 3 weeks × 3 cycles; gemcitabine 1000 mg/m2 day 1, 8 + cisplatin 80 mg/m2 day 1) followed by intensity-modulated radiotherapy (IMRT; 70 Gy, 33 fractions, 5 fractions/week, 1 fraction/day) alone. PD-1 blockade toripalimab (240 mg per cycle) will start on day 1 of the first cycle IC and continue every 3 weeks for 6 cycles till the end of IMRT, involving the whole-course of IC + IMRT alone. The first and last 3 cycles of toripalimab are administrated concurrently with IC and IMRT, respectively. After 3 weeks of the completion of IMRT, adjuvant toripalimab (240 mg per cycle) will begin every 3 weeks for 11 cycles.
  Interventions: Drug: PD-1 blocking antibody; Drug: Gemcitabine; Drug: Cisplatin (80mg/m2); Radiation: Intensity-modulated radiotherapy
- Toripalimab Combined with Induction Chemotherapy Followed by Concurrent Chemoradiotherapy (Active Comparator): All participants will receive induction chemotherapy (IC; every 3 weeks × 3 cycles of gemcitabine 1000 mg/m2 day 1, 8 + cisplatin 80 mg/m2 day 1) followed by concurrent chemoradiotherapy (CCRT; every 3 weeks × 2 cycles of cisplatin + IMRT 70 Gy, 33 fractions, 5 fractions/week, 1 fraction/day). PD-1 blockade toripalimab (240 mg per cycle) will start on day 1 of the first cycle IC and continue every 3 weeks for 6 cycles till the end of CCRT, involving the whole-course of IC + CCRT. The first and last 3 cycles of toripalimab are administrated concurrently with IC and CCRT, respectively. After 3 weeks of the completion of CCRT, adjuvant toripalimab (240 mg per cycle) will begin every 3 weeks for 11 cycles.
  Interventions: Drug: PD-1 blocking antibody; Drug: Gemcitabine; Drug: Cisplatin (80mg/m2); Drug: Cisplatin (100mg/m2); Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: PD-1 blocking antibody — 1. IC phase of PD-1 blocking antibody: every 3 weeks × 3 cycles; 240 mg, day 1; start on day 1 of the first cycle IC and continue every 3 weeks for 3 cycles till the end of IC.
  2. IMRT phase of PD-1 blocking antibody: every 3 weeks × 3 cycles; 240 mg, day 1; start on day 1 of IMRT or CCRT and continue every 3 weeks for 3 cycles till the end of IMRT.
  3. Adjuvant PD-1 blocking antibody: every 3 weeks × 11 cycles; 240 mg, day 1
  Other Names: PD-1 Blockade
Drug: Gemcitabine — Gemcitabine as induction chemotherapy, 1000 mg/m2 day 1, 8 per cycle, every 3 weeks for 3 cycles
  Other Names: GEM
Drug: Cisplatin (80mg/m2) — Cisplatin as induction chemotherapy, 80 mg/m2 day 1 per cycle, every 3 weeks for 3 cycles
  Other Names: DDP
Drug: Cisplatin (100mg/m2) — Cisplatin as concurrent chemotherapy, 100 mg/m2 day 1 per cycle, every 3 weeks for 2 cycles
  Other Names: DDP
  Arms: Toripalimab Combined with Induction Chemotherapy Followed by Concurrent Chemoradiotherapy
Radiation: Intensity-modulated radiotherapy — Definitive IMRT of 70 Gy, 33 fractions, 5 fractions/week, 1 fraction/day
  Other Names: IMRT

SUMMARY:
This is a phase 3, multi-center, randomized controlled trial, with the purpose to evaluate the therapeutic efficacy and safety of PD-1 blockade (toripalimab) combined with the de-intensified chemoradiotherapy sparing concurrent cisplatin (i.e., toripalimab incorporated into induction chemotherapy and radiotherapy) in high-risk locoregionally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This phase 3, multi-center, randomized controlled trial plans to enroll 532 patients with newly-diagnosed, pathologically-proven, untreated locoregionally advanced nasopharyngeal carcinoma (LANPC) at high-risk of distant metastasis (T4N1 and T1-4N2-3, according to American Joint Committee on Cancer [AJCC]/Union for International Cancer Control [UICC] 8th edition clinical staging system). Patients will receive 3 cycles of induction chemotherapy (IC; gemcitabine-cisplatin regimen) followed by 1) experimental arm (de-intensification group): intensity-modulated radiotherapy (IMRT) alone or 2) control arm (standard group): 2 cycles of concurrent cisplatin plus IMRT (CCRT). For both of the two arms, toripalimab will be adopted on day 1 of the first cycle IC and continue every 3 weeks for 6 cycles till the end of IMRT, with the first and last 3 cycles of toripalimab administrated along with IC and CCRT/IMRT, respectively. After three weeks of the completion of IMRT, adjuvant toripalimab will be used every 3 weeks for 11 cycles, and therefore the entire treatment process is expected to last for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65;
2. Pathological type: non-keratinizing carcinoma (World Health Organization criteria);
3. Diagnosed with LANPC (T4N1, T1-4N2-3) according to the 8th edition clinical staging system of the American Joint Committee on Cancer [AJCC]/Union for International Cancer Control [UICC];
4. ECOG performance score: 0 to 1;
5. Normal bone marrow function: white blood cell count > 4×109/L, hemoglobin > 90g/L, platelet count > 100×109/L;
6. Normal values of thyroid function, amylase and lipase examination, pituitary function, inflammation and infection indicators, myocardial enzymes, and ECG results. For patients older than 50 years with a smoking history, normal lung function are required. Patients with abnormal ECG and/or a history of vascular disease (but not meeting the exclusion criteria listed in the exclusion criteria 7) need further testing and require normal results of myocardial function and color Doppler ultrasound.
7. Normal liver and kidney function: total bilirubin ≤ 1.5 × upper limit of normal (ULN); alanine transaminase and aspartate transaminase ≤ 2.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; creatinine clearance rate ≥ 60 ml/min;
8. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule;
9. Subjects with pregnancy ability must agree to use reliable contraceptive measures from screening to 1 year after treatment.

Exclusion Criteria:

1. Hepatitis B virus surface antigen (HBsAg) positive and HBV DNA > 1×10E3 copies/ml; anti-hepatitis C virus positive;
2. Anti-human immunodeficiency virus (HIV) positive or diagnosed with acquired immune deficiency syndrome (AIDS);
3. Active tuberculosis: active tuberculosis in the past 1 year should be excluded regardless with treatment; history of active tuberculosis over 1 year should be excluded except that previous regulatory anti-tuberculosis treatment is proved;
4. Active, known or suspected autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, pituitary, nephritis, vasculitis, hyperthyroidism, hypothyroidism and asthma requiring bronchiectasis). Exceptions are type I diabetes mellitus, hypothyroidism requiring hormone replacement therapy, skin disorders requiring no systemic treatment (such as vitiligo, psoriasis or alopecia);
5. Previous interstitial lung disease or pneumonia requiring oral or intravenous steroid therapy;
6. Chronic treatment with systemic glucocorticoid (dose equivalent to or over 10 mg prednisone per day) or any other form of immunosuppressive therapy. Subjects who used inhaled or topical corticosteroids were eligible;
7. Uncontrolled heart disease, for example: 1) heart failure (NYHA level ≥ 2); 2) unstable angina; 3) myocardial infarction in past 1 year; 4) supraventricular or ventricular arrhythmia requiring treatment or intervention;
8. Pregnant or lactating women (pregnancy test should be considered for women with sexual life and fertility);
9. Previous or concurrent with other malignant tumors, except for adequately treated non-melanoma skin cancer, cervical carcinoma in situ and thyroid papillary cancer;
10. Allergy to macromolecular protein preparations, or any component of nivolumab;
11. Active infection requiring systemic treatment;
12. Receiving live vaccine within 30 days of the initial nivolumab;
13. History of organ transplantation;
14. History of psychotropic disease, alcoholism or drug abuse; other situation assessed by the investigators that may compromise the safety or compliance of patients, such as serious disease requiring timely treatment (including mental illness), severe laboratory abnormalities, or family-social risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3-year
  Failure-free survival is measured from day of diagnosis until treatment failure, death from any cause, or last follow-up visit, whichever occurred first
Incidence rate of all-grade vomiting | Through study completion, an average of 1 year
  Incidence rate of all-grade vomiting during treatment assessed by clinicians according to the Common Terminology Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
Overall survival (OS) | 3-year
  Overall survival is measured from day of diagnosis until death due to any cause or the latest known date alive
Locoregional failure-free survival (LRFFS) | 3-year
  Locoregional failure-free survival is measured from day of diagnosis until local or regional recurrence
Distant failure-free survival (DFFS) | 3-year
  Distant failure-free survival is measured from day of diagnosis until distant metastasis
Incidence rate of investigator-reported adverse events (AEs) | 3-year
  Analysis of investigator-reported adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
Incidence rate of patient-reported adverse events (AEs) | 3-year
  Analysis of patient-reported adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by patients themselves
Quality of life (QoL): questionnaire | week 1, 20, 40, 64
  Changes in QoL of participants from initial treatment to 6 months after the completion of 6 cycles adjuvant PD-1 blocking antibody. QoL is evaluated with the use of (1) the head-and-neck-specific module (H&N35) of the Quality of Life Questionnaire-Core 30 module (QLQ-C30), which is established by European Organization for Research and Treatment of Cancer (EORTC) and (2) the general and head-and-neck-specific module of the evaluation tool developed by the Functional Assessment of Cancer Therapy (FACT). Scores for the module range of H&N35 QLQ-C30 from 0 to 100, with higher scores indicating better functioning or well-being or higher symptom burden (scales measuring symptom burden were reverse-scored to facilitate presentation)
Tumor response | Through study completion, an average of 1 year
  Evaluation of tumor response (CR, PR, SD, PD, NA) performed after induction chemotherapy, radiotherapy, and adjuvant PD-1 immunotherapy.

OTHER OUTCOMES:
Correlation between pre-treatment PD-L1 expression level and FFS | 3-year
  Pre-treatment PD-L1 expression level of tumor cell is evaluated centrally by means of immunohistochemical testing. This is a single assessment with only one unit of measure, since the correlation is aimed to be roughly categorized into positive and negative.
Correlation between pre-treatment PD-L1 expression level and OS | 3-year
  Pre-treatment PD-L1 expression level of tumor cell is evaluated centrally by means of immunohistochemical testing. This is a single assessment with only one unit of measure, since the correlation is aimed to be roughly categorized into positive and negative.
Correlation between the percentage of tumor-infiltrating lymphocytes (TILs) and PFS | 3-year
  TILs are lymphoid cells (T cells) that infiltrate solid tumors (intra-tumoral TILs) and stroma (stromal TILs), which play an important role in the tumor microenvironment. This is a single assessment with only one unit of measure, since the correlation is aimed to be roughly categorized into positive and negative.
Correlation between the percentage of tumor-infiltrating lymphocytes (TILs) and OS | 3-year
  TILs are lymphoid cells (T cells) that infiltrate solid tumors (intra-tumoral TILs) and stroma (stromal TILs), which play an important role in the tumor microenvironment. This is a single assessment with only one unit of measure, since the correlation is aimed to be roughly categorized into positive and negative.
Evaluate failure-free survival in the subgroup of age at diagnosis (year) | 3-year
  Subgroup analysis
Evaluate failure-free survival in the subgroup of gender (male and female) | 3-year
  Subgroup analysis
Evaluate failure-free survival in the subgroup of plasma Epstein-Barr virus DNA level | 3-year
  Subgroup analysis
Evaluate failure-free survival in the subgroup of clinical stage | 3-year
  Subgroup analysis
Evaluate the regression of tumor and parotid glands during radiotherapy | From the first fraction of radiotherapy to the end of treatment
  Evaluate the anatomical (size, volume, and 3-dimensional axis) and dosimetric changes of primary tumor, lymph node, and parotid glands during 33-fractionation radiotherapy by using cone beam computed tomography
Failure-free survival 2 (FFS 2) | within 10 years
  The time from randomization to the second or subsequent disease progression after the initiation of new anticancer therapy, or death from any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Principal Investigator — Sun Yat-sen University
Locations (12):
- China (12):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - First People's Hospital of Foshan, Foshan, Guangdong
  - Panyu central hospital, Guangzhou, Guangdong
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hubei Province Cancer Hosiptal, Wuhan, Hubei
  - Tongji Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangxi Province Cancer Hospital, Nanchang, Jiangxi
  - Zhejiang Province Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Result] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Result] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Result] Fang W, Yang Y, Ma Y, Hong S, Lin L, He X, Xiong J, Li P, Zhao H, Huang Y, Zhang Y, Chen L, Zhou N, Zhao Y, Hou X, Yang Q, Zhang L. Camrelizumab (SHR-1210) alone or in combination with gemcitabine plus cisplatin for nasopharyngeal carcinoma: results from two single-arm, phase 1 trials. Lancet Oncol. 2018 Oct;19(10):1338-1350. doi: 10.1016/S1470-2045(18)30495-9. Epub 2018 Sep 10. PMID 30213452
- [Result] Wang FH, Wei XL, Feng J, Li Q, Xu N, Hu XC, Liao W, Jiang Y, Lin XY, Zhang QY, Yuan XL, Huang HX, Chen Y, Dai GH, Shi JH, Shen L, Yang SJ, Shu YQ, Liu YP, Wang W, Wu H, Feng H, Yao S, Xu RH. Efficacy, Safety, and Correlative Biomarkers of Toripalimab in Previously Treated Recurrent or Metastatic Nasopharyngeal Carcinoma: A Phase II Clinical Trial (POLARIS-02). J Clin Oncol. 2021 Mar 1;39(7):704-712. doi: 10.1200/JCO.20.02712. Epub 2021 Jan 25. PMID 33492986
- [Derived] DIAMOND Study Group; Xu C, Liang XY, Huang XQ, Jin F, Yang KY, Hu GY, Zhu XD, Wang Y, Huang Y, Zhang N, Hu DS, Guo L, Zou GR, Chen XZ, Xiao SW, Li JG, Shen LF, Li YY, Huang J, Long GX, Li L, Huang L, She LJ, Wu Y, Zeng WH, Qiang MY, Liu WX, Su Y, Tang LL, Xie FY, Han F, Lu LX, Xiang YQ, Mao YP, Li WF, Liu X, Yang Q, Zhou GQ, Guo R, Ouyang PY, Wang XH, Chen L, Liu LT, Lin L, Li JB, Lin AH, Zhao HY, Hong SB, Jie YS, Huang HL, Tang XH, Zeng YC, Yun JP, Zang SB, Du ZM, Ye ZL, Liu LZ, Tian L, Li HJ, Peng YL, Liu N, Li YQ, Liang YL, Wei HM, Chen YP, Zhang Y, Du XJ, Lv JW, Sun Y, Ma J. Toripalimab Combination Therapy Without Concurrent Cisplatin for Nasopharyngeal Carcinoma: The DIAMOND Randomized Clinical Trial. JAMA. 2025 Sep 16;334(11):973-983. doi: 10.1001/jama.2025.13205. PMID 40839372